CLINICAL TRIAL: NCT05523245
Title: Predicting the Efficacy of Neoadjuvant Therapy in Patients With Locally Advanced Rectal Cancer Using an AI Platform Based on Multi-parametric MRI
Acronym: DLARC
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital of Jinan University (Other)
Responsible Party: Principal Investigator, xiaochun meng, The Director of Diagnostic Radiology Department, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2021ZSLYEC-478
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2024-10

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- complete response: Patients receiving neoadjuvant therapy achieved pathological complete response before LARC.
- non complete response: Patients receiving neoadjuvant therapy did not achieve pathological complete response before LARC.

SUMMARY:
Establish a deep learning model based on multi-parameter magnetic resonance imaging to predict the efficacy of neoadjuvant therapy for locally advanced rectal cancer.This study intends to combine DCE with conventional MRI images for DL, establish a multi-parameter MRI model for predicting the efficacy of CRT, and compare it with the DL and non-artificial quantitative MRI diagnostic model constructed by conventional MRI to evaluate the role of DL in MRI predicting CRT. And this study also tries to build a DL platform to assess the efficacy of LARC neoadjuvant radiotherapy and chemotherapy, accurately assess patients' complete respose (pCR) after CRT, and provide an important basis for guiding clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion or colonoscopic pathology of rectal cancer
* Age over 18 years
* Informed consent and signed informed consent form

Exclusion Criteria:

* Poor magnetic resonance image quality, such as severe artifacts
* Previous treatment for rectal cancer
* History or combination of other malignant tumours
* Not Locally Advanced Rectal Cancer (LARC)
* Not received neoadjuvant therapy or not completed neoadjuvant therapy
* No surgery
* Time interval between MRI and surgery was more than 2 weeks
* Patients were lost to follow-up and voluntarily withdrew from the study due to adverse reactions or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer (LARC) treated with neoadjuvant therapy and radical surgery
Sampling Method: Non-Probability Sample
Enrollment: 1700 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of models in prediction tumor response | baseline and pre-operation
  The area under curve (AUC) of Receiver Operating Characteristic (ROC) curves of models in identifying the pCR candidates from non-pCR individuals among neoadjuvant therapy treated LARC patients will be calculated.

SECONDARY OUTCOMES:
The specificity of models in prediction tumor response | baseline and pre-operation
  The sensitivity of models in identifying the pCR candidates from non-pCR individuals among neoadjuvant therapy treated LARC patients will be calculated.
The sensitivity of models in prediction tumor response | baseline and pre-operation
  The sensitivity of models in identifying the pCR candidates from non-pCR individuals among neoadjuvant therapy treated LARC patients will be calculated.
The positive predictive value of models in prediction tumor response | baseline and pre-operation
  The positive predictive value of models in identifying the pCR candidates from non-pCR individuals among neoadjuvant therapy treated LARC patients will be calculated.
The negative predictive value of models in prediction tumor response | baseline and pre-operation
  The negative predictive value of models in identifying the pCR candidates from non-pCR individuals among neoadjuvant therapy treated LARC patients will be calculated.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong